CLINICAL TRIAL: NCT06183307
Title: Effects of Nattokinase on Inflammation and Cardiovascular Risk Markers in Patients With Dyslipidemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: Denise Mafra17
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Diseases; Dyslipidemias; Inflammation
Keywords: nattokinase; Cardiovascular Diseases; Inflammation; fibrinogen
MeSH Terms: conditions — Cardiovascular Diseases; Dyslipidemias; Inflammation | interventions — nattokinase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nattokinase group (Experimental): Participants will receive 1 capsule per day, providing the active nattokinase daily, at a dosage of 100mg, standardized at 2,000 Fibrinolytic Units.
  Interventions: Dietary Supplement: Nattokinase
- Placebo Group (Placebo Comparator): The placebo group will receive the same amount of 100mg placebo, at the same time, containing corn starch.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nattokinase — Participants will receive 1 capsule per day, providing the active nattokinase daily, at a dosage of 100mg, standardized at 2,000 Fibrinolytic Units for 2 months
  Arms: Nattokinase group
Dietary Supplement: Placebo — The placebo group will receive 1 capsule per day with 100mg containing corn starch for 2 months.
  Arms: Placebo Group

SUMMARY:
The study aims to evaluate the effect of the nattokinase enzyme on inflammation and markers of cardiovascular risk in participants with dyslipidemia. A longitudinal double-blind randomized clinical trial will be carried out, involving hypertensive participants with dyslipidemia for two months.

DETAILED DESCRIPTION:
Nattokinase has potent fibrinolytic/antithrombotic, antihypertensive, antiatherosclerotic, lipid-lowering, antiplatelet/anticoagulant and neuroprotective activities. Nattokinase is capable of inhibiting platelet aggregation by blocking the formation of thromboxane and inactivating the type 1 plasminogen activator inhibitory factor. Recently, it was proposed that nattokinase can attenuate oxidative stress and the inflammatory process in in vitro and animal models. However, there are no studies in dyslipidemic patients evaluating these data.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes;
* Over 18 years of age;
* Isolated increase in LDL-c (LDL-c ≥ 160 mg/dL);
* Isolated increase in triglycerides (TG ≥ 150 mg/dL or ≥ 175 mg/dL, without fasting);
* increased LDL-c (LDL-c ≥ 160 mg/dL)
* TG (TG ≥ 150 mg/dL or ≥ 175 mg/dL, without fasting);
* Reduction in HDL-c (men < 40 mg/dL and women < 50 mg/dL) alone or in association with an increase in LDL-c or TG. If TG ≥ 400 mg/dL.
* Individuals who are already using lipid-lowering therapy (statins or non-statins) will also be included.

Exclusion Criteria:

* Participants with autoimmune and infectious diseases, diabetes, cancer and AIDS;
* Pregnant women;
* Participants using catabolic drugs or antibiotics
* Participants on anticoagulant medication
* Participants using antioxidant vitamin supplements, prebiotic, probiotic or synbiotic and who are allergic to corn or soy starch.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-08-03 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change of inflammatory status in the participants | Baseline and 8 weeks
  Get blood samples to evaluate the supplementation effects in inflammatory biomarkers: interleukin 6 (IL-6), tumor necrosis factor-alpha (TNF-alpha), C-reactive protein (CRP).

SECONDARY OUTCOMES:
Change in plasma fibrinogen levels, lipid peroxidation and improvement in lipid profile. | Baseline and 8 weeks
  Get blood samples to evaluate the supplementation effects in plasma fibrinogen, lipid profile (HDL-c, LDL-c, total cholesterol) and lipid peroxidation.

CONTACTS AND LOCATIONS:
Overall Officials: Ludmila Cardozo, PhD, Principal Investigator — Universidade Federal Fluminense
Locations (1):
- Denise Mafra, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No
Participant data will not be public to other research unless necessary.